CLINICAL TRIAL: NCT03135223
Title: Development of Intervention Strategies to Increase Physical Activity and Reduce Sedentary Behaviour in Secondary Schoolgirls by Means of Participatory Health Research
Brief Title: Participatory Research to Promote Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Principal Investigator, Vakgroepsport, Prof. Greet Cardon, University Ghent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWO13/PDO/191
Record Dates: First submitted 2017-04-18; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Health Behavior
Keywords: Physical activity
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: One intervention and one control condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Co-created, school-based intervention to promote physical activity
  Interventions: Behavioral: Co-created intervention to promote physical activity
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Co-created intervention to promote physical activity — A working group of girls and researcher co-created a school-specific intervention to promote physical activity
  Arms: Intervention group

SUMMARY:
Secondary schoolgirls have the most unhealthy profile regarding physical activity and sedentary behaviour of all age groups. Since both behaviours independently contribute to various health outcomes, an effective intervention to promote physical activity and to reduce sedentary behaviour needs to be developed.

Many interventions fail to induce changes in health behaviour, as they often use a top-down approach with limited input from the end-users (i.e. the secondary schoolgirls) of the intervention programmes. This project uses a participatory health research approach by actively involving the girls in the entire research process. A co-creation group was set up per intervention school (n=3), including girls and a researcher which co-created a school-specific intervention, tailored to the needs and interests of those girls.

The effect of participatory process were evaluated via a clustered randomized controlled trial using an intervention and control condition and a pre- and post-test design. Effects on physical activity and related determinants (e.g. self-efficacy, attitude, etcetera) were evaluated. The hypothesis was that girls from the intervention condition would improve their physical activity levels and related determinants compared to no changes among girls from the control schools. The process was evaluated as well using focus group research and the hypothesis was that girls who participate in the co-creation groups would be positive about the process and will feel empowered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, female pupils of secondary schools (aim: 10th grade) who volunteer to participate in the study

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 196 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Increase in the mean overall physical activity level of adolescent girls | one schoolyear
  Overall physical activity (expressed in average minutes per day) is calculated by summing active transportation (i.e. minutes spent in active transportation to school and in leisure time per day) and sport participation (i.e. minutes spent in physical education, extra-curricular sports or physical activities at school and during leisure time per day), measured by the reliable and valid Flemish Physical Activity Questionnaire.

SECONDARY OUTCOMES:
Increase in the mean value of determinants related to physical activity | one schoolyear
  Three individual (i.e. self-efficacy, perceived benefits and perceived barriers) and six sociocultural determinants (i.e. peer and parental modelling, peer and parental co-participation and peer and parental encouragement) were assessed using questions from previous studies examining adolescents' health behaviour, of which the predictive validity and reliability have been demonstrated previously. Three school-related determinants (i.e. relationship with classmates, involvement in organising school activities and relationship with teachers) were assessed using items from the Flemish Health Behaviour in School-aged Children questionnaire.